CLINICAL TRIAL: NCT05561218
Title: Dispersion of Shoulder Helical Axes Before and After Physical Therapy in Patients With Shoulder Instability
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: CLF21/02
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Shoulder Instability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Shoulder instability is associated with neuromuscular control alterations. Helical Axes (HAs) dispersion is influenced by joint morphology and neuromuscular control and its analysis can be used to quantify the Center of Rotation (CoR) displacement.

The aim of the study is to evaluate the effects of an exercise-based training on shoulder HAs dispersion during upper limb movements in patients with shoulder instability and to assess the association between shoulder arthrokinematics and instability-related symptoms.

25 patients with shoulder instability and 25 healthy subjects (aged between 18 and 50) will be enrolled. The HAs dispersion will be assessed during the performance of two upper limb task, shoulder flexion and shoulder rotation. Kinematics will be recorded by an optoelectronic system and HAs dispersion was computed using Mean Distance (MD) and Mean Angle (MA).

Pain and functional impairments will be assesed through the DASH scale, NRS scale, simple shoulder test (SST). Quality of life will be assessed with SF-12 scale.

Outcomes measures will be evaluated at the enrolment (T0), after one week (T1), after 12 weeks (T2) and after one month (T3). Between T1 and T2 patients perform a 12 weeks home-based exercise protocol and 12 outpatient physical therapy sessions.

DETAILED DESCRIPTION:
This will be a single center, observational study that will be conducted in Humanitas Research Hospital.

Patients with symptomatic shoulder instability be enrolled. An orthopaedic surgeon will confirm the diagnosis and recruit patient.

Age-matched heathy subjects, without history of shoulder pain or trauma in the last year, will be enrolled in the study.

Patients will perform a 12 weeks home exercise protocol (5 sessions of 15-20 minutes per week). The exercise-based treatment will be in line with the current literature and will focus on gaining neuromuscular control in different biomechanical contexts.

The home-based training will be divided in 5 different stages. In line with previous studies, the first phase will comprise isometric contractions that aim to the activation of the shoulder muscles and enhance their synergy. The second phase will include closed kinetic chain exercises to enhance physiological neuromuscular activation and shoulder functional stability, as previous studies suggested. The third phase will be a progression of phase 2 since it will use more challenging closed kinetic chain exercises .During phase four, patient will do closed kinetic chain exercises and low-load open kinetic chain exercises. During the fifth phase will include open kinetic chain and task-oriented exercises. Patients will attend one outpatient physical therapy session every week supervised by a physical therapist, who will show the exercises of the following week. Patient will also have a leaflet that will describe in detail each exercise.

Treatment compliance will be tracked every week through a diary in which patients have to report exercises performed.

HAs dispersion, measured during shoulder flexion and shoulder rotation, will be quantified through the parameters of mean distance (MD) and mean angle (MA). MD describes displacement of HAs, providing a measure of CoR movement, whereas MA describes orientation of HAs, showing the ability to perform a movement on a single plane of motion [3-9]. Kinematics will be recorded by optoelectronic system (BTS SMART-DX, Spa), consisting of 8 optical cameras with a sampling frequency of 100 Hz.

Some retro-reflective markers will be positioned on the trunk and upper limb, in particular a cluster of 5 markers on the posterolateral surface of the arm and 6 other markers on the following landmarks: C7, T8, jugular notch, xiphoid process, ulnar styloid and acromial angle.

Pain and functional impairments will be assesed through the DASH scale, NRS scale, simple shoulder test (SST). Quality of life will be assessed with SF-12 scale.

Patient will be evaluated at the enrolment (T0), after one week (T1), at the end of the training of 12 weeks (T2) and after one month from the end of the training (T3). During this last month patient will be asked to stop exercising.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* Positivity to (at least) one of the three tests described in literature to asses multidirectional shoulder instability: sulcus sign, drawer test and apprehension test
* First episode of glenohumeral dislocation or subluxation treated with assisted reduction
* Presence of anatomical damage compatible with conservative treatment
* Presence of pain or apprehension in the last month

Exclusion Criteria:

* Subjects requiring surgical glenohumeral stabilization
* History of shoulder surgery
* Medically unstable subjects who, at the time of inclusion, have a neurological, internal or musculoskeletal disease that could affect functional or motor recovery

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Patients will be enrolled among Humanitas Hospital outpatients
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Helical Axes (HAs) dispersion analysis | At baseline, after 1 week, after 12 weeks of training and at 1 month after the training end.
  Changes in HAs dispersion to quantify the displacement of Center of Rotation during upper limb movements was quantified through parameters of MD and MA, which represent HAs displacement and orientation. HAs analysis will be performed through an optoelectronic system (BTS SMART-DX, Spa), consisting of 8 optical cameras and retroreflective markers.

SECONDARY OUTCOMES:
Numeric pain rating scale (0- best outcome, 100 worst outcome) | At baseline, after 12 weeks of training and at 1 month after the training end.
  Changes in shoulder pain
Disability Arm Shoulder Hand (0- best outcome, 100 worst outcome) | At baseline, after 12 weeks of training and at 1 month after the training end.
  Changes in shoulder function
Simple shoulder test (0- worst outcome, 12 best outcome) | At baseline, after 12 weeks of training and at 1 month after the training end.
  Changes in shoulder function
Short form - 12 items (12- best outcome, 57 worst outcome) | At baseline, after 12 weeks of training and at 1 month after the training end.
  Changes in quality of life